CLINICAL TRIAL: NCT04290195
Title: Safety and Efficacy of Ziv Aflibercept in Myopic Choroidal Neovascularisation ,Central Retinal Vein Occlusion and Resistant Diabetic Macular Edema
Brief Title: Use of Ziv Aflibercept in Different Retinal Diseases
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Amin El Sayed Nawar (Other)
Collaborators: Tanta University (Other)
Responsible Party: Sponsor-Investigator, Amin El Sayed Nawar, Amin Nawar MD.Lecturer of Ophthalmology, Tanta University
Organization: Tanta University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2AA
Record Dates: First submitted 2020-02-23; First posted 2020-02-28 (Actual); Last update posted 2021-10-11 (Actual); Status verified 2021-10

CONDITIONS: Central Retinal Vein Occlusion With Macular Edema
Keywords: myopic choroidal neovascularisation
MeSH Terms: interventions — aflibercept

STUDY DESIGN:
Intervention Model Description: Resistant diabetic macular edema,non ischaemic central retinal vein occlusion and myopic choroidal neovascularisation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- ziv aflibercept patients (Experimental): 20 eyes of myopic CNV,20 eyes with resistant diabetic macular edema and 15 eyes with non ischaemic CRVO
  Interventions: Drug: Ziv-Aflibercept 25 MG/ML [Zaltrap]

INTERVENTIONS:
Drug: Ziv-Aflibercept 25 MG/ML [Zaltrap] — Intravitreal injection of 1.25 mg of ziv aflibercept in patients
  Other Names: zaltrap

SUMMARY:
A prospective interventional case series study was conducted on 20 eyes of 20 patients with active myopic choroidal neovascularisation (CNV) ,20 eyes with resistant diabetic macular edema and 15 eyes with non ischaemic central retinal vein occlusion(CRVO) after approval of the Ethical Committee of the Faculty of Medicine, Tanta University . All procedures were carried out under the tenets of the Helsinki Declaration. Written consent was provided by all participants after discussing the procedure, alternative treatment plans, follow-up schedules, and possible benefits and risks.

DETAILED DESCRIPTION:
Intravitreal injection of 1.25 mg of ziv aflibercept was done in different retinal diseases including myopic CVN,resistant diabetic macular edema to previous ranibizumab injection and non ischaemic CRVO .Thorough ophthalmic evaluation was done including BCVA(best corrected visual acuity) ,anterior and posterior segment examination ,fundus fluorescein angiography and OCT(optical coherence tomography) were performed for all patients .Injection was repeated as PRN(pro re nata) method after one month if persistent intraretinal or subretinal fluid was found.

ELIGIBILITY:
Inclusion Criteria:

* The study included treatment naive patients suffering from recently diagnosed active myopic subfoveal or juxtafoveal CNV less than 2 months documented by fundus fluorescein angiography (FFA)and optical coherence tomography (OCT ) , pathological myopia more than 6 D was included .

Exclusion Criteria:

* Previous intraocular surgery .
* Coincident retinal pathology as diabetic retinopathy, retinal vein occlusion .
* CNV due to other causes like age related macular degeneration ,angioid streaks,trauma and choroiditis.
* Extrafoveal myopic CNV .
* Patients received other lines of treatment for CNV like photodynamic therapy ,laser photocoagulation or intravitreal injection of triamcinolone or other anti VEGF(vascular endothelial growth factor) agents.
* Known glaucoma , clinical suspicion of glaucoma or IOP(intraocular pressure) more than 20 mmHg.
* Prior ocular inflammation.
* The presence of retinal degeneration.
* Patients who didnot complete 6 months of follow up

Ages: 31 Years to 63 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 55 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2020-01-01 (Actual)

PRIMARY OUTCOMES:
Improvement of BCVA by log MAR(minimum angle of resolution) and reduction of CMT after intravitreal injection | 6 months
  To assess sustained improvement of BCVA(Best corrected visual acuity) and reduction of the CMT (central macular thickness) after intravitreal injection of zivaflibercept

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University, Tanta, El Gharbia, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Chan WM, Ohji M, Lai TY, Liu DT, Tano Y, Lam DS. Choroidal neovascularisation in pathological myopia: an update in management. Br J Ophthalmol. 2005 Nov;89(11):1522-8. doi: 10.1136/bjo.2005.074716. PMID 16234465
- [Derived] Nawar AE, Wasfy T, Shafik HM. Switching to ziv-aflibercept in resistant diabetic macular edema non responsive to ranibizumab injection. BMC Ophthalmol. 2022 Jun 29;22(1):287. doi: 10.1186/s12886-022-02503-x. PMID 35768859
- [Derived] Nawar AE, Shafik HM. Pilot study of ziv-aflibercept in myopic choroidal neovascularisation patients. BMC Ophthalmol. 2020 Oct 19;20(1):414. doi: 10.1186/s12886-020-01679-4. PMID 33076864
- See also: medical journal that contains multiple papers — http://www.ncbi.nlm.nih.gov